CLINICAL TRIAL: NCT04770844
Title: Development of a Developmental Prognostic Tool for the Premature Child Based on Automated Spontaneous Motor Analysis
Acronym: AGMA
Status: Terminated | Type: Observational
Why Stopped: inclusion difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other); Laboratoire EA SNA=EPIS 4607. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20CH234; 2020-A03335-34 (Other: ANSM)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Premature Birth
Keywords: premature children; motor skill; developmental prognostic; prognostic tool
MeSH Terms: conditions — Premature Birth | interventions — Health Facility Merger

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- premature child: 300 premature child will be included. They will have three acquisitions during hospitalization.
  Interventions: Other: Acquisitions

INTERVENTIONS:
Other: Acquisitions — Three acquisitions of 1 hours during hospitalization will be realized:
  * a few days after hospitalization,
  * in the middle of the hospitalization,
  * a few days before hospital discharge. The child will be lying on his back in a heated cradle and filmed with a specific camera. The signal will be obtained by 2k ZED 2 stereo camera in order to obtain a three-dimensional location of the child

SUMMARY:
Prematurity is a major risk factor for poor neurodevelopmental outcomes. The clinical and neuroradiological evaluations proposed during the neonatal period to assess the developmental prognosis of children born prematurely are not sensitive and nor specific. The analysis of spontaneous motor activity by Prechtl's method has a better predictive value but is currently unfeasible in clinical routine. The study's principal objective is to describe the standardized values of complexity, variability, and fluidity of general movements.

ELIGIBILITY:
Inclusion Criteria:

* Birth before 33 week of amenorrhea;
* Hospitalization in the Neonatal Department of the Saint-Étienne University Hospital
* Patient affiliated or entitled to a social security scheme;
* Authorization to shoot the holders of parental authority;
* Consent to participate in the study by the holders of parental authority

Exclusion Criteria:

* Need for ventilatory support;
* Difficulty of thermal regulation contraindicating the use of a heating cradle;
* Refusal of authorization to shoot by holders of parental authority;
* Refusal of participation in the study of holders of parental authority.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children borned before 33 week of amenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Automatized quantification of complexity of general movements (spatial variation). | Year: 3
  Measured by analyze of all acquisitions.
Automatized quantification of variability of general movements (temporal variations) | Year: 3
  Measured by analyze of all acquisitions.
Automatized quantification of fluidity of general movements (uniform distribution) | Year: 3
  Measured by analyze of all acquisitions.

SECONDARY OUTCOMES:
Comparison between our quantitative analysis and qualitative analysis according to the reference method of Pretchl | Year: 3
  Measured by analyze of all acquisitions.

CONTACTS AND LOCATIONS:
Overall Officials: ANTOINE GIRAUD, MD, Principal Investigator — CHU ST ETIENNE FRANCE
Locations (1):
- Chu de St Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No